CLINICAL TRIAL: NCT03663647
Title: Multicentral Retrospective Chart Review Study of Targeted Therapy Use in Patients With BRAF V600 Advanced (Unresectable or Metastatic) Cutaneous Melanoma in Routine Clinical Practice in Russian Federation
Brief Title: Advanced Melanoma in Russian Experience
Acronym: ADMIRE
Status: Completed | Type: Observational
Sponsor: MelanomaPRO, Russia (Other)
Collaborators: Crocus Medical B.V. (Unknown)
Responsible Party: Principal Investigator, Kristina Orlova, MD, PhD, Senior Сlinical Researcher, MelanomaPRO, Russia
Other Study IDs: ADMIRE
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Cutaneous Melanoma, Stage IV; BRAF V600 Mutation
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective chart review Study of patients with BRAF V600 positive advanced (unresectable or metastatic) melanoma, who were treated with targeted therapy in routine clinical practice in Russian Federation

DETAILED DESCRIPTION:
This study is an observational multicentral retrospective chart review study in patients with BRAF V600 positive advanced (unresectable or metastatic) cutaneous melanoma, who have treated by BRAF inhibitors (BRAFi) or MEK inhibitors (MEKi) in routine clinical practice in Russia. 300 patients will be included in the study.

The study does not aim to prove any formal hypothesis and does not imply any intervention in standard medical care, and all medical events recorded during the study have already occurred. The data sources of this study will be medical records, patients' charts and other related medical documentation that allows to fully follow the course of the disease and collect all the necessary information according to Protocol.

For identification of molecular genetic markers that cause resistance and sensitivity to targeted therapy, an analysis of tumor tissue will be provided in the laboratory of biological microchips "Institute of Molecular Biology. V.A. Engelhardt" of the Russian Academy of Sciences. The analyzed materials will be paraffin blocks with samples of tumor tissue of only patients with primary resistance to targeted therapy (inhibitors BRAF / +/- MEK inhibitor).

In the course of the study, the Contract Research Organization (CRO) "Crocus Medical B.V." will conduct periodic monitoring visits to ensure that the data collected are accurate and credible. Regular monitoring visits include Source Data Verification (SDV) in accordance with the monitoring plan, monitoring compliance with the research procedures, as well as the proper and timely maintenance of the main clinical study documents, including the reporting provided for by the rules of good clinical practice, the legislation of the Russian Federation and Standard Operating Procedures (SOPs) of the CRO.

The investigators will be responsible for the collection and provision of all clinical and laboratory data, as well as safety data, that are entered in electronic Case Report Forms (e-CRF), and must ensure data authenticity and compliance with the primary documentation.

Before hard database lock, the database will be inspected in order to reveal missing and suspicious data. The queries will be generated to correct or fill-in such data. In case the data failed to refine, their will be considered as missing, no data-imputation methods are planned.

One of the efficacy endpoints of the study is defined as overall survival which represents the time-to-event data, these data will be analyzed with Kaplan-Meyer method and Cox regression. Time to event will be defined as a number of days passed from start of treatment until any-cause death. Patients alive until the end of study will be right-censored by the end-of-study day or by the day of preliminary withdrawal. Based on Kaplan-Meyer curves the following parameters would be accessed: median survival, one- and two-year survival. The Cox regression will include the following covariates: age, sex, baseline therapy, presence of metastasis in brain, baseline level of lactic dehydrogenase (LDH), number of tissues with metastasis, time from the beginning of the target therapy, etc. Additional covariates could be also accessed when necessary. The hazard ratio (HR) along with 95% confidence interval will be evaluated for each covariate.

Analyses of categorical efficacy endpoints (number of patients taken different therapies, objective response rate, number of patients with molecular genetics alterations) will be performed with chi-square criterion or Fisher's exact test in case of any expected frequencies below 5. In addition, the logistic regression could be build based on the above mentioned covariates. The odds ratio (OR) along with 95% confidence interval will be evaluated for each covariate.

The progression-free survival (PFS) will be analyzed analogously as described above for the overall survival data. Time to event will be defined as a number of days passed from treatment start until either any-cause death or documented disease progression whichever occurs first. Patients without event will be right-censored by the end-of-study day or by the day of preliminary withdrawal. Based on Kaplan-Meyer curves the following parameters would be accessed for all the patients as well as for the subgroups of baseline therapy (target therapy, immunochemistry, chemotherapy): 6-, 12-, 18- and 24-months progression-free survival. In addition, the PFS will be analyzed for the patients treated with BRAFi as a monotherapy with successive inclusion of the MEKi.

Time to response and duration of response data will be analyzed similarly. Time to response will be defined as a number of days passed from treatment start until first documented response to the therapy. Non-responders will be right-censored by the end-of-study day or by the day of preliminary withdrawal. This analyses will be conducted for all the patients as well as for the subgroups of baseline therapy (target therapy, immunochemistry, chemotherapy).

Analyses of the duration of response will be performed only among the responders. Duration of the response will be defined as a number of days passed from the first documented response until either any-cause death or documented disease progression whichever occurs first. Patients responding until the study end will be right censored by the end-of-study day or by the day of preliminary withdrawal.

The data on duration of the therapy will be presented with descriptive statistics for each therapy line.

Adverse events (AE) and Serious Adverse Events (SAE) will be coded according to MedDRA. Each AE/SAE will be summarized with counts and frequencies. The data on AE will be tabulated by System Organ Classes (SOC) and presented with indication their preferred terms (PT) by baseline therapy and severity. When necessary, the comparison of frequencies of AEs/SAEs between subgroups will performed with chi-square criterion or Fisher's exact test in case of any expected frequencies below 5.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmed cutaneous melanoma
* BRAF V600 mutation
* Treated by at least one therapy line including BRAFi / MEKi

Exclusion Criteria:

* No data of targeted therapy usage and treatment outcomes (data of evaluation of effect and data of objective examination)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with BRAF V600 advanced (unresectable or metastatic) cutaneous melanoma, who were treated by BRAFi or MEKi in routine clinical practice in Russian Federation
Sampling Method: Non-Probability Sample
Enrollment: 382 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2019-04-27 (Actual); Study Completion 2019-04-27 (Actual)

PRIMARY OUTCOMES:
Approach to therapy in patients with metastatic or unresectable BRAF mutant melanoma | 4 years
  Percentages of patients who were treated by targeted, immunotherapy and chemotherapy or other therapy types of treatment usage in each line of treatment

SECONDARY OUTCOMES:
Overall survival (OS) of patients with stage III (unresectable) and stage IV BRAF V600-positive cutaneous melanoma | 5 years
  The median OS of patients with unresectable advanced BRAF mutant melanoma during targeted therapy
Overall survival (OS) of patients with stage III (unresectable) and stage IV BRAF V600-positive cutaneous melanoma | 5 years
  2 year OS rate of patients with unresectable advanced BRAF mutant melanoma during targeted therapy
The response rate during therapy in patients with unresectable advanced BRAF mutant melanoma | 4 years
  The ORR by subgroup of patients with unresectable advanced BRAF mutant melanoma during targeted therapy
Disease control rate (DCR) in patients with unresectable advanced BRAF mutant melanoma | 4 years
  The DCR by subgroup of patients with unresectable advanced BRAF mutant melanoma
Progression free survival (PFS) of patients with stage III (unresectable) and stage IV BRAF V600-positive cutaneous melanoma | 4 years
  The median PFS and 24 months PFS rate of patients with unresectable advanced BRAF mutant melanoma during targeted therapy
The incidence of adverse events during targeted therapy | 5 years
  The rate of all grade and grade 3-5 adverse events and the rate of discontinuation of study drug(s) due to adverse events.
The PFS in patients with advanced BRAF mutant melanoma during targeted therapy by type of BRAF mutation | 4 years
  The PFS rate according to the mutation BRAF subtype
The OS in patients with advanced BRAF mutant melanoma during targeted therapy by type of BRAF mutation | 4 years
  The OS rate according to the mutation BRAF subtype

OTHER OUTCOMES:
Frequency of occurrence of any progression types on different treatments | 4 years
  The rate of progression and type according to TNM classification for melanoma

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Orlova, MD, PhD, Study Chair — Association Professional Melanoma Society (MELANOMA.PRO)
Locations (11):
- Russia (11):
  - Moscow Regional Oncologic Dispensary, Balashikha
  - Belgorod Oncologic Dispensary, Belgorod
  - Republican Clinical Oncologic Dispensary, Cheboksary
  - Kaluga Regional Clinical Oncologic Dispensary, Kaluga
  - N.N. Blokhin National Medical Research Centre of Oncology, Moscow
  - Clinical Oncologic Dispensary, Omsk
  - City Clinical Oncologic Dispensary, Saint Petersburg
  - N.N. Petrov National Medical Research Centre of Oncology, Saint Petersburg
  - St. Petersburg Clinical Scientific and Practical Center for Specialized Types of Medical Care (Oncology), Saint Petersburg
  - Tula Regional Oncologic Dispensary, Tula
  - Voronezh Regional Clinical Oncologic Dispensary, Voronezh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Orlova KV, Ledin EV, Zhukova NV, Orlova RV, Karabina EV, Volkonskiy MV, Stroyakovskiy DL, Yurchenkov AN, Protsenko SA, Novik AV, Vorotilina LV, Moiseenko FV, Chang VL, Kazmin AI, Tkachenko SA, Gamaunov SV, Naskhletashvili DR, Samoylenko IV, Vikhrova AS, Utyashev IA, Kharkevich GY, Petenko NN, Shubina IZ, Demidov LV. Real-World Experience with Targeted Therapy in BRAF Mutant Advanced Melanoma Patients: Results from a Multicenter Retrospective Observational Study Advanced Melanoma in Russia (Experience) (ADMIRE). Cancers (Basel). 2021 May 21;13(11):2529. doi: 10.3390/cancers13112529. PMID 34064013
- See also: Real-World Experience with Targeted Therapy in BRAF Mutant Advanced Melanoma Patients: Results from a Multicenter Retrospective Observational Study Advanced Melanoma in Russia (Experience) (ADMIRE) — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC8196785/